CLINICAL TRIAL: NCT04393623
Title: Understanding and Targeting Stress Reactivity in Women Veterans With Alcohol Misuse
Brief Title: Stress, Emotion Regulation, and Alcohol in Women Veterans
Acronym: SERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MHBB-017-18F; DVA/CSR&D CDA-2 CX001951 (Other Grant/Funding Number: Veterans Health Administration, Office of Research)
Record Dates: First submitted 2020-04-27; First posted 2020-05-19 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Use Disorder; Post Traumatic Stress Disorder
Keywords: Alcohol Use Disorder; Women Veterans; Endocrinology; Cognitive Reappraisal; Microintervention; Progesterone; Posttraumatic Stress Disorder; Psychophysiology; Heart Rate Variability
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be urn randomized to either an experimental (cognitive reappraisal) or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Reappraisal Microintervention (Experimental): The CR microintervention (session 1) is drawn from Barlow & colleagues empirically supported treatment for emotional disorders (the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders). The microintervention consist of four sections: (1) Introduction to cognitive appraisal; (2) Introducing the idea of "thinking traps" that prevent reappraisal and maintain negative emotion; (3) Describing cognitive reappraisal as a strategy that can help the participant "get out" of such thinking traps; (4) Providing an example of this process (situation> negative appraisal > negative emotion > thinking trap > opportunity for cognitive reappraisal) and have participants provide a personalized example.
  Interventions: Behavioral: Cognitive Reappraisal
- Psychoeducation (Control) (Active Comparator): The manualized psychoeducational control module, serving as an attentional control, is derived from two sources: 1. The first session of the Women's Health Education Manual, which provides psychoeducation about the basic body systems and their function, with focus on components of the immune system and 2. Fact sheets published by the American College of Obstetricians and Gynecologists(ACOG), providing female-specific facts about cancer and heart health. None of this psychoeducation discusses potential relevancy of alcohol use, nor will any behavior changes be suggested during the control microintervention.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive Reappraisal — This cognitive reappraisal microintervention lasts 45-60 minutes.
  Arms: Cognitive Reappraisal Microintervention
Behavioral: Psychoeducation — This psychoeducational microintervention lasts 45-60 minutes.
  Arms: Psychoeducation (Control)

SUMMARY:
The purpose of the study "Stress, Emotion Regulation, and Alcohol in Women Veterans" is to learn about the effects of negative emotion and stress on behavior (including alcohol use) among women Veterans, including women with and without posttraumatic stress disorder. Additionally, the study looks at whether a woman's use of emotion regulation techniques changes the association between stress or negative emotion and behavior. Lastly, the study examines how women's reactions to stress, and the effects of stress, vary across the menstrual cycle - depending on the level of circulating hormones.

DETAILED DESCRIPTION:
Aims for the current study are two-fold: 1. conduct a randomized trial testing the effects of an emotion regulation skill (cognitive reappraisal) on stress-induced drinking among women with alcohol misuse and varying levels of co-occurring PTSD; 2. examine whether progesterone levels and/or severity of co-occurring PTSD - factors which impact women's stress reactivity and emotion regulation - moderate the effectiveness of the cognitive reappraisal in reducing stress-induced drinking.

The proposed study will combine experimental, in-person sessions with daily self-report data from the Veterans to assess the effect of cognitive reappraisal on alcohol craving, cognitive (inhibitory) control, physiological arousal (HRV), and alcohol use. Participation will take place across a period of at least 35 days, to encompass an entire menstrual cycle. All participants complete all sections of the study - the experimental sessions and the longitudinal (35-day) data collection.

ELIGIBILITY:
Inclusion Criteria:

* Current alcohol misuse, defined as scoring 3 or higher on the AUDIT-C
* If using other illicit substances, alcohol is their primary substance of use
* Alcohol use in the past 45 days
* Able to write and speak in English
* Served in the U.S. Military
* Willing to provide blood samples at laboratory sessions to assay hormone levels and take urine ovulation tests at home

Exclusion Criteria:

* Psychotic symptoms or uncontrolled Bipolar Disorder (screened for during session 1 using SCID-5 screening modules)
* Brain damage or were in an accident that affects ability to complete the computerized task
* Current (past 3 months) active suicidal ideation or intent
* Current pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 81 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Alcohol Craving during Experimental Sessions | Two separate days during the study (ie. on two of the study days, which last up to 75 days)
  Craving will be measured via the Alcohol Craving Questionnaire - Short Form (ACQ-SF). The ACQ-SF comprises 12 items and is used to assess alcohol cravings among alcohol users in the current moment. Participants are asked to rate how much they agree or disagree with each statement, each regarding how they feel or think about alcohol in the moment. Each item is scored on a 7-point Likert scale that reflects their agreement on a scale of "strongly disagree" to "strongly agree".
Change in Inhibitory Control during Experimental Sessions | Two separate days during the study (ie. on two of the study days, which last up to 75 days)
  Inhibitory Control, a measure of behavioral impulsivity, will be assessed with a computerized task (a stop-signal task, STOP-IT). Participants' stop signal reaction time (SSRT) reflects varying levels of inhibitory control (lower SSRT reflects better inhibitory control).
Change in Heart Rate Variability (HRV) during Experimental Sessions | Two separate days during the study (ie. on two of the study days, which last up to 75 days)
  Heart rate variability (HRV), a physiological measure of arousal and shown to be a measure of stress reactivity and impacted by successful emotion regulation, will be assessed with a Biopac MP160 data acquisition unit with an ECG amplifier that allows for the measurement of HRV.
Change in frequency of alcohol use prior to and through study completion | Retrospectively for 45 days prior to study enrollment, and through study completion (up to 75 days post-baseline)
  The Alcohol Timeline Follow Back (TLFB) assesses frequency/quantity of drinking. The TLFB will be used at all laboratory sessions to fill in any potentially missing data from the daily logs

SECONDARY OUTCOMES:
Change in intensity of daily negative affect | Daily, through study completion (up to 75 days post-baseline)
  The Positive and Negative Affect Schedule (PANAS) is a 10 item questionnaire that measures self reported positive and negative affect. Each item is rated on a 5-point scale of 1 (not at all) to 5 (very much). Scores range from 10-50.
Change in depression symptoms from baseline to study completion, un to 75 days | Baseline, end of study (up to 75 days)
  Beck Depression Inventory II (BDI-II) is a self-report questionnaire assessing depression symptoms over the prior two weeks (scores range 0-63) and higher scores indicate greater depression symptomatology. All item scores are summed to attain a total score.
Change in depression symptoms from baseline to study completion, un to 75 days | Baseline, end of study (up to 75 days)
  PTSD Checklist for DSM-5 with Life Events checklist and Criterion A (PCL-5) is a 20-item self-report questionnaires assessing current symptoms of PTSD, used to assess current (past 30 days) PTSD severity. Total scores are calculated by summing all values. Scores on the PCL-5 range from 0-80 and reflect a global PTSD severity score, with higher scores indicating greater severity.
Change in use of adaptive and maladaptive emotion regulation strategies | weekly, through study completion (up to 75 days post-baseline)
  Emotion Regulation Questionnaire (ERQ) is 10-item questionnaire measuring emotion regulation. Items are rated on a 7-point Likert-scale ranging from 1 (strongly disagree) to 7 (strongly agree). Specifically, the measure assesses use of the strategies cognitive reappraisal and emotional suppression, which are separate subscales. Higher scores reflect greater use of each type of emotion regulation strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Cathryn Glanton Holzhauer, PhD, Principal Investigator — VA Central Western Massachusetts Healthcare System, Leeds, MA
Locations (1):
- VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT04393623/ICF_000.pdf